CLINICAL TRIAL: NCT01352286
Title: A Phase I/IIa, Dual-cohort, Two-site, Clinical Trial Evaluating the Safety and Activity of Redirected Autologous T Cells Expressing a High Affinity TCR Specific for NY-ESO-1 Administered Post ASCT in Patients With Advanced Myeloma
Brief Title: Redirected Auto T Cells for Advanced Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209393; ADP 01411 (Other: Adaptimmune Therapeutics)
Record Dates: First submitted 2011-05-04; First posted 2011-05-11 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Received initial treatment previously; Autologous stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous Genetically modified T cells (Experimental): Patients with advanced myeloma and who are candidates for autologous stem cell transplants, or syngeneic stem cell transplants (SSCT), will be eligible. Prior to full screening on this study, patients will undergo prescreening to evaluate HLA-A type and presence of NY-ESO-1c259T/LAGE antigen. Patients will undergo a steady-state mononuclear cell apheresis for T cell collection, with an optional second collection. Once mononuclear cells have been collected, patients (or donors in the case of SSCT) will then undergo hematopoietic stem cell mobilization. Patients will receive a dose >0.1-1 x 10¹º anti-CD3/anti-CD28-costimulated autologous T cells which have been genetically modified to express high affinity NY-ESO-1c259 TCRs.
  Interventions: Genetic: Autologous Genetically modified T cells

INTERVENTIONS:
Genetic: Autologous Genetically modified T cells — Patients will undergo myeloma restaging at days +42, +100, 6 months, 9 months and 1 year post infusion. At this point, in accordance with FDA Guidelines, all patients will enter long term follow up (LTFU) and be followed biannually for monitoring for gene transfer delayed adverse events until year 5 post infusion. From year 5, all patients will require annual LTFU visits for monitoring for delayed adverse events until year 15 after receiving the genetically modified T cells.
  Patients whose disease progresses prior to year 1 will enter LTFU at time of progression; however these patients will be seen quarterly from progression until year 1 post infusion and then follow the LTFU schedule mentioned above.

SUMMARY:
The purpose of this study is to 1) evaluate the safety and tolerability of autologous genetically modified T cells transduced to express the high affinity NY-ESO-1c259 TCR in HLA-A2+ subjects and 2) measure the incidence of GVHD in patients following infusion of TCR modified autologous T cells.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of autologous genetically modified T cells. Genetic material is transferred into the subject's previously harvested autologous T cells to redirect them to target myeloma cells rather than their usual target. Study subjects must have systemic or multifocal myeloma requiring autologous stem cell transplantation whose disease has relapsed or incompletely responded to prior therapy or have high-risk features. Subjects must also have measureable disease on study entry, as defined by quantifiable or detectable levels of serum or urine paraprotein or elevated serum free light chains with an abnormal ratio.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma has relapsed, progressed, or failed to respond after at least one prior course of therapy (consisting of at least 2 treatment cycles or months of therapy)
* Myeloma has responded partially to initial therapy but a complete response (immunofixation negative and normal serum free light chain) has NOT developed after a minimum of 3 cycles or months of initial therapy
* Myeloma has high-risk features as defined by the presence of one or more cytogenetic abnormalities known to confer a poor outcome even after standard auto-transplants: complex karyotype (≥ to 3 abnormalities), t(4;14), t(14;16), del (17) (p13.1), and/or chromosome 13 abnormalities. These patients may be enrolled even while in complete or near-complete remission
* Measurable disease on study entry, as defined by quantifiable or detectable levels of serum or urine paraprotein or elevated serum free light chains with abnormal ratio
* Patients who are in complete remission at the time of proposed study entry (serum and urine immunofixation consistently negative and normal serum free light chains) are not eligible unless their disease meets the criteria for high-risk as defined in protocol
* Ages 18-80
* ECOG performance status 0-2 (unless due solely to bone pain)
* Prior to Lenalidomide maintenance phase, all study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®
* Females subjects of childbearing potential must have a negative pregnancy test and both male and female (of childbearing potential) subjects must agree to use reliable methods of contraception during the study.
* Lenalidomide treatment phase: able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin)
* HLA-A201 patients must have confirmed expression of NY-ESO-1 and/or LAGE. HLA-A2 patients must have the A-201 allele

Adequate vital organ function as defined below:

* Serum creatinine ≤3.0 mg/dl and not on dialysis
* WBC at least 3000/mm³, platelet count at least 100,000/mm³
* SGOT ≤ to 2 x upper limit of normal and bilirubin ≤ to 2.0 mg/dl (unless due to Gilbert's syndrome)
* Left ventricular ejection fraction (LVEF) ≥ 45%. A lower LVEF is permissible if a formal cardiologic evaluation reveals no evidence for clinically significant functional impairment
* Adequate pulmonary function with mechanical parameters ≥ 40% predicted (FEV1, FVC, TLC, DLCO). Patients who are unable to complete PFTs due to bone pain or fracture must have a high resolution CT scan of the chest and must have acceptable arterial blood gases defined as a room air PO2 greater than 70 mmHg
* Patients should have recovered from any toxicities related to prior therapy or at least returned to their baseline level of organ function.
* Patients should be off of glucocorticoids for at least 2 weeks and/or other therapies for at least 1 week prior to enrollment

Exclusion Criteria:

* Pregnant or nursing females
* HIV or HTLV-1/2 seropositivity
* History of myelodysplasia
* History of chronic active hepatitis or liver cirrhosis (if suspected by laboratory studies, should be confirmed by liver biopsy)
* Active Hepatitis B (as defined by positive Hepatitis B surface antigen); positive Hepatitis C virus (HCV) antibody is NOT an exclusion
* Prior allogeneic transplant
* History of severe autoimmune disease requiring steroids or other immunosuppressive treatments
* Active immune mediated diseases including: connective tissue diseases, uveitis, sarcoidosis, inflammatory bowel disease, multiple sclerosis
* Evidence or history of other significant cardiac, hepatic, renal, ophthalmologic, psychiatric, or gastrointestinal disease which would likely increase the risks of participating in the study
* Active bacterial, viral, or fungal infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05-13 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20063

REFERENCES:
- [Background] Stadtmauer EA, Faitg TH, Lowther DE, Badros AZ, Chagin K, Dengel K, Iyengar M, Melchiori L, Navenot JM, Norry E, Trivedi T, Wang R, Binder GK, Amado R, Rapoport AP. Long-term safety and activity of NY-ESO-1 SPEAR T cells after autologous stem cell transplant for myeloma. Blood Adv. 2019 Jul 9;3(13):2022-2034. doi: 10.1182/bloodadvances.2019000194. PMID 31289029

RESULTS

PARTICIPANT FLOW:
Groups:
- NYESO-1ᶜ²⁵⁹T Cells Administered Intravenously: Participants who received lentivirus-mediated genetically engineered NYESO-1ᶜ²⁵⁹T following autologous stem cell transplantation (ASCT)
Period: Overall Study
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells Administered Intravenously
Started | 25
Received T-cells | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who received NY-ESO-1ᶜ²⁵⁹T following ASCT
Groups:
- NYESO-1ᶜ²⁵⁹T Cells: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 59 [45 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Related to Study Treatment
Description: Number of Participants with Adverse Events related to study treatment
Time Frame: Day -40 to Year 1 post-treatment
Population: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT
Measure: Number; unit: participants
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
Number analyzed (Participants) | 25
participants | 24

2. Secondary Outcome: Number of Participants With Response Per International Myeloma Working Group (IMWG) 2011 Criteria
Description: Objective Response Rate (ORR) of sCR (stringent complete response), CR (complete response), VGPR (very good partial response), PR (partial response)
Time Frame: Change from Baseline at Day 42, 100, 180, 270 and Year 1
Population: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT
Measure: Count of Participants; unit: Participants
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
Number analyzed (Participants) | 25
Participants
  Day 42 | 20
  Day 100 | 19
  Day 180 | 16
  Day 270 | 13
  Year 1 | 11

3. Secondary Outcome: Best Objective Response (BOR)
Description: Number of participants with Best Objective Response of sCR, CR, VGPR, or PR
Time Frame: Best Objective Response prior to initiation of lenalidomide and at Year 1
Population: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT with Best Objective Response (BOR) data.
Measure: Count of Participants; unit: Participants
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
Number analyzed (Participants) | 25
Participants
  Prior to Initiation of Lenalidomide : sCR | 1
  Prior to Initiation of Lenalidomide : CR | 0
  Prior to Initiation of Lenalidomide : VGPR | 12
  Prior to Initiation of Lenalidomide : PR | 7
  Year 1 : sCR | 2
  Year 1 : CR | 1
  Year 1 : VGPR | 13
  Year 1 : PR | 5

4. Secondary Outcome: Duration of Response (DOR), Progression Free Survival (PFS), Overall Survival (OS)
Description: Calculated median DOR, PFS, OS
Time Frame: DOR: Initial date of response to date of progressive disease or death PFS: Date of first T -cell infusion to earliest date of disease progression of death due to any cause OS: Date of first T-cell infusion to date of death from any cause.
Population: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT
Measure: Median (95% Confidence Interval); unit: median months
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
Number analyzed (Participants) | 25
median months
  DOR | 12.2 [7.6 to 29.8]
  PFS | 13.5 [8.9 to 31.1]
  OS | 35.1 [22.7 to NA] — The 95% upper confidence limits for median overall survival could not be calculated because of the high number/proportion (11 participants/44%) of participants alive at the time of the analysis.

5. Secondary Outcome: Peak Persistence of Modified T-cells in the Peripheral Blood
Description: Measurement of NY-ESO-1ᶜ²⁵⁹T cells in blood
Time Frame: Post-infusion through Day 42
Population: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT
Measure: Mean (Full Range); unit: copies per μg of DNA
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
Number analyzed (Participants) | 25
copies per μg of DNA | 143728.793 [7560.10 to 284312.37]

6. Secondary Outcome: Marrow Antigen Expression Pre-and Post-infusion
Description: Number of participants with NY-ESO-1 and LAGE or LAGE-1a expression in the marrow post-infusion
Time Frame: Pre- and post-infusion
Population: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT with expression data at all points.
Measure: Number; unit: participants
Groups:
- NYESO-1ᶜ²⁵⁹T Cells: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT with data at pre-and post-infusion time points
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
Number analyzed (Participants) | 25
participants
  Day 100 : NY-ESO-1 | 16
  Day 100 : LAGE or LAGE-1a | 16
  Day 180 : NY-ESO-1 | 14
  Day 180 : LAGE or LAGE-1a | 14

7. Secondary Outcome: Engraftment of Gene-modified Pentamer+ CD4+ T Cells and CD8+ T Cells
Description: Number of participants with engraftment in blood and bone marrow
Time Frame: Post Treatment
Population: Participants who received NYESO-1ᶜ²⁵⁹T following ASCT with engraftment data.
Measure: Number; unit: participants
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
Number analyzed (Participants) | 25
participants
  CD4+ : Blood | 11
  CD4+ : Bone Marrow | 11
  CD8+ : Blood | 11
  CD8+ : Bone Marrow | 11

ADVERSE EVENTS:
Time Frame: Day -40 to Year 1 post-treatment
Description: Participants who received NY-ESO-1ᶜ²⁵⁹T following ASCT
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells
All-Cause Mortality (participants affected / at risk) | 14/25
Serious Adverse Events (participants affected / at risk) | 17/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NYESO-1ᶜ²⁵⁹T Cells (N=25)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Graft versus host disease (Immune system disorders) | 2 (2)
Hypoxia (Gastrointestinal disorders) | 2 (2)
Staphylococcal infection (Infections and infestations) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ejection Fraction (Investigations) | 1 (1)
Failure to Thrive (Metabolism and nutrition disorders) | 1 (1)
Graft versus host disease in gastrointestinal tract (Gastrointestinal disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Myoglobin blood (Investigations) | 1 (1)
Myoglobin urine (Investigations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NYESO-1ᶜ²⁵⁹T Cells (N=25)
Nausea (Gastrointestinal disorders) | 25 (25)
Anaemia (Blood and lymphatic system disorders) | 24 (24)
Diarrhea (Gastrointestinal disorders) | 24 (24)
Decreased appetite (Metabolism and nutrition disorders) | 23 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (18)
Platelet count decreased (Investigations) | 12 (12)
Fatigue (General disorders) | 22 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 (20)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Pyrexia (General disorders) | 20 (20)
Hypokalemia (Metabolism and nutrition disorders) | 19 (19)
Vomiting (Gastrointestinal disorders) | 19 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
WBC decreased (Investigations) | 13 (13)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
Neutrophil count decreased (Investigations) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Hypocalcaemia (Metabolism and nutrition disorders) | 14 (14)
Oedema peripheral (General disorders) | 14 (14)
Stomatitis (Gastrointestinal disorders) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 13 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Constipation (Gastrointestinal disorders) | 12 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 (12)
Hypophosphataemia (Metabolism and nutrition disorders) | 12 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 (12)
Headache (Nervous system disorders) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 11 (11)
Chills (General disorders) | 10 (10)
Hypotension (Vascular disorders) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (8)
Insomnia (Psychiatric disorders) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7)
Oral Pain (Gastrointestinal disorders) | 7 (7)
Pain (General disorders) | 7 (7)
Alanine aminotransferase increased (Investigations) | 6 (6)
Anxiety (Psychiatric disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Dizziness (Nervous system disorders) | 6 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Tachycardia (Cardiac disorders) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 5 (5)
Candida infection (Infections and infestations) | 5 (5)
Graft Versus Host Disease (GVHD) (Immune system disorders) | 4 (4)
Localized edema (General disorders) | 5 (5)
Lymphocyte count decreased (Investigations) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood creatinine increased (Investigations) | 4 (4)
Depression (Psychiatric disorders) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Herpes zoster (Infections and infestations) | 4 (4)
Hypertension (Vascular disorders) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
Mucosal inflammation (General disorders) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Oesophagitis (Gastrointestinal disorders) | 4 (4)
Paresthesia (Nervous system disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Weight decreased (Investigations) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Autoimmune disorder (Immune system disorders) | 3 (3)
Blood creatinine decreased (Investigations) | 3 (3)
Catheter site pain (General disorders) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 3 (3)
Confusional state (Psychiatric disorders) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3)
Malaise (General disorders) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neuralgia (Nervous system disorders) | 3 (3)
Neutropenic colitis (Gastrointestinal disorders) | 3 (3)
Oral candidiasis (Infections and infestations) | 3 (3)
Oral dysaesthesia (Gastrointestinal disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tremor (Nervous system disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Abdominal tenderness (Gastrointestinal disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Catheter site discharge (General disorders) | 2 (2)
Catheter site hemorrhage (General disorders) | 2 (2)
Chest discomfort (General disorders) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Delirium (Psychiatric disorders) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Face edema (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Flushing (Vascular disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (2)
International normalized ratio increased (Investigations) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Peripheral swelling (General disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Scab (Skin and subcutaneous tissue disorders) | 2 (2)
Sinus headache (Nervous system disorders) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Staphylococcal infection (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Vision blurred (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT01352286/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT01352286/SAP_001.pdf